CLINICAL TRIAL: NCT01367015
Title: A Randomized Clinical Trial on Comparison of Early Versus Late Initiation of Feeding in Preterm Small for Gestation Infants Below 35 Weeks Gestation With Prenatal Absent or Reversal of End Diastolic Flow (AREDF) in Umbilical Artery
Brief Title: Early Versus Late Initiation of Feeding in Premature Growth Restricted Newborns With Absent or Reversed End Diastolic Flow On Umbilical Artery Doppler (AREDF)
Acronym: AREDF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Collaborators: Sir Ganga Ram Hospital (Other); Maulana Azad Medical College (Other); Vardhman Mahavir Medical College And Safdarjung Hospital (Other); Fernandez Hospital (Unknown)
Responsible Party: Dr Sushma Nangia, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: A-20/ April 2006
Record Dates: First submitted 2011-06-01; First posted 2011-06-06 (Estimated); Last update posted 2011-06-06 (Estimated); Status verified 2006-04

CONDITIONS: Prematurity of Fetus; Postnatal Growth Disorder
Keywords: Preterm; SGA; AREDF; Early feeding; Late feeding; Feed intolerance; Necrotizing enterocolitis; Days to achieve Full Feeds defined as 150 mL/kg
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Feeding (Experimental): Early feeding group received minimal enteral feed (MEF) of 8 ml/kg of expressed human milk of the biologic mother for 48 hours after randomization followed by regular feeding with feed increments of 20ml/kg/day to reach 150 ml/kg.
  Interventions: Other: Early Feeding
- Late feeding (Active Comparator): Late feeding group was kept NPO for a period of 48 hours after randomization followed by minimal enteral feed (MEF) of 8 ml/kg of expressed human milk of the biologic mother for 48 hours and thereafter received regular feeding with feed increments of 20ml/kg/day till full enteral feeds of 150 ml/kg/day were achieved
  Interventions: Other: Late Feeding

INTERVENTIONS:
Other: Early Feeding — Feeding with expressed breast milk @ 8ml/kg/day for 48 hrs after randomization at 60+/-12 hrs of life
  Arms: Early Feeding
Other: Late Feeding — Nil per oral for another 48 hrs after randomization at 60+/-12 hrs of life followed by Feeding with expressed breast milk @ 8ml/kg/day for 48 hrs
  Arms: Late feeding

SUMMARY:
The purpose of the study is to compare early versus late initiation of enteral feeding in premature growth restricted babies below the gestational age of 35 weeks born to mothers with prenatal absent or reversal of end diastolic flow in the umbilical artery. Normally the blood flow from the mother to the baby brings all the nutrients required for growth and the very vital oxygen required for survival. These deprived babies with poor blood flow adapt to the not so conducive uterine environment by certain adjustments in blood supply to internal organs. This permits the best possible blood flow to brain heart etc., which are the vital organs and whose adequate functioning is required for survival. As a consequence, the gut (intestines) gets poor blood supply and hence its appropriate functioning may be jeopardized. Such 'premature growth restricted' babies are at increased risk of further growth faltering if not fed adequately as also to a condition called 'Necrotising enterocolitis' if fed liberally like other healthy neonates, characterized by abdominal distension, blood in stools and inability to feed for longer durations thereby further affecting growth. In the past such babies (after birth) were not fed for days together which compromised their growth even further. It is not clear whether continuing to withhold feeds for prolonged duration will prevent NEC but lead to growth faltering and initiating feeds early will potentiate NEC with further compromised growth and increased morbidity. There are no randomized trials on feeding strategies in this group of neonates and hence the investigators planned to carry out this study on comparison of early versus delayed initiation of feeding in preterm SGA infants with AREDF.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm neonates below 35 weeks gestation born at the study center(s)
2. Small for gestational age (SGA) ie weight < 10th centile for gestation
3. Absent or reverse end diastolic flow (AREDF) in umbilical artery

Exclusion Criteria:

1. Babies with major congenital malformations.
2. Babies with severe asphyxia as defined by apgar score <4 at 5 min of life with cord/within one hour of life pH< 7.0.
3. Shock requiring pressor support at the time of randomization.
4. Babies born with gastrointestinal surgical conditions precluding enteral feeding.
5. Babies with abdominal distension, bilious or hemorrhagic aspirates or recurrent vomiting at the time of randomization.
6. Refusal to obtain consent.
7. Gestation below 26 weeks.
8. Hydrops fetalis.

Ages: 48 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Days to achieve full feeds defined as 150mL/kg | upto 12 weeks (84 days)
  First day of the three days when full enteral feeding of 150 ml/kg has been achieved and sustained as recorded from the nursing chart of the neonate

SECONDARY OUTCOMES:
Days to regain birth weight | upto 16 weeks (112 days)
  After the initial fall in weight the first day when birth weight is regained or crossed and the value remains above the birth weight for subsequent 2 days will be recorded as day of life birth weight has been regained.
Feed intolerance | 12 weeks (84 days)
  Feed intolerance was measured as number of episodes of any of the following symptoms per infant till he/she reached full feeds of 150ml/kg and sustained it for 2 days.
  * bilious or hemorrhagic aspirates( irrespective of the volume),
  * vomiting ( >2 times in 12 hours duration) and
  * clear or milky aspirate >50% of the previous feed volume necessitating feed stoppage for 24 hours
Duration of stay | 12 - 16 weeks (84 - 112 days)
  This was taken to be the interval between birth and the day the newborn was discharged home.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sushma Nangia, MBBS, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Dr Sushma, New Delhi, National Capital Territory of Delhi, India